CLINICAL TRIAL: NCT03708237
Title: Effectiveness of Ropinirole and Gabapentin for the Treatment of Restless Legs Syndrom in Patients on Maintenance Hemodialysis: a Randomized, Blinded, Placebo-Controlled Trial
Brief Title: Effectiveness of Ropinirole and Gabapentin for the Treatment of RLS in Patients on Maintenance HD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment suspended due to COVID-19 pandemic and will not resume.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00084427
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2021-06

CONDITIONS: Restless Legs Syndrome; End Stage Renal Disease
MeSH Terms: conditions — Restless Legs Syndrome; Kidney Failure, Chronic | interventions — ropinirole; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebos (Placebo Comparator): Placebo Dose: Not Applicable Route: Mouth Regimen: Daily 2 hours before bed Duration: 6 months
  Interventions: Drug: Placebos
- Ropinirole (Experimental): Drug: ropinirole Dose: 0.25 - 2 mg as tolerated Route: Mouth Regimen: Daily 2 hours before bed Duration: 6 months
  Interventions: Drug: Ropinirole
- Gabapentin (Experimental): Drug: gabapentin Dose: 100 - 300 mg as tolerated Route: Mouth Regimen: Daily 2 hours before bed Duration: 6 months
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Ropinirole — ROPINIROLE has been approved by Health Canada for the treatment of idiopathic Parkinson's disease. Immediate release ropinirole is an orally administered non-ergoline dopamine agonist that is extensively metabolized by the liver. Ropinirole has not been approved by Health Canada for the treatment of moderate to severe RLS.
  Other Names: ACT-ROPINIROLE
  Arms: Ropinirole
Drug: Gabapentin — GABAPENTIN has been approved by Health Canada for the management of epilepsy. Immediate release gabapentin is an orally administered anticonvulsant primarily excreted through the kidneys. Gabapentin has not been approved by Health Canada for the treatment of moderate to severe RLS.
  Other Names: APO-GABAPENTIN
  Arms: Gabapentin
Drug: Placebos — Opaque gel capsules filled with methylcellulose 1500 filler
  Arms: Placebos

SUMMARY:
Restless legs syndrome (RLS) is a neurologic disorder characterized by 1) an urge to move the legs, 2) uncomfortable sensations in the legs, 3) symptoms that are often worse the evening or when at rest , and 4) may be temporarily relieved by physical activity.

The overall prevalence of RLS in the general population is estimated to be around 10%, however, it is significantly in the end stage kidney disease (ESKD) population is significantly higher (approximately 30%). Studies have shown that RLS has a substantial negative impact on both the physical and the mental health dimensions of quality of life (QOL), such as depression, anxiety, pain, fatigue and sleep disorder.

While non-pharmacological treatments should be considered for all patients, pharmacological management of RLS is indicated when the affects patient's sleep or quality of life. Gabapentin and dopamine agonists such as ropinirole are usually the first choices in treating RSL. Although these medications are also used in patients with renal impairment, few studies provide treatment data for the hemodialysis population. Treatment recommendations for this population are largely based on data obtained in the general population.

This study aims to evaluate effectiveness of ropinirole and gabapentin for the treatment of restless legs syndrome in patients on maintenance hemodialysis.

DETAILED DESCRIPTION:
Purpose

Restless legs syndrome (RLS), also known as Willis-Eskbom disease, is a neurologic disorder characterized by 1) an urge to move the legs, 2) uncomfortable sensations in the legs, 3) symptoms that are often worse the evening or when at rest , and 4) may be temporarily relieved by physical activity. While the precise pathogenic mechanisms responsible for uremic RLS remain unknown, there is evidence to support involvement of dopaminergic dysfunction and reduced iron stores.

RLS is separated into primary/idiopathic and secondary forms. Secondary RLS is usually associated with underlying medical conditions such as end-stage kidney disease (ESKD). The overall prevalence of RLS in the general population is estimated to be around 10%. However, the prevalence of RLS in the ESKD population is significantly higher. A systematic review calculated weighted mean RLS prevalence of 30% (range: 8-52%) in ESKD. Studies have shown that RLS has a substantial negative impact on both the physical and the mental health dimensions of quality of life (QOL), such as depression, anxiety, pain, fatigue and sleep disorder.

While non-pharmacological measure should be considered for all patients, pharmacological treatment for RLS is indicated when the symptoms lead to significant insomnia or impaired quality of life. Although only two medications have been approved by Health Canada, there is a long list of medications that have been used in management of RLS symptoms. Gabapentin and dopamine agonists are usually the first choices in treating RSL. Although marketed in Canada, gabapentin and ropinirole have not been approved by Health Canada for the treatment of moderate-severe restless legs sydnrome.

Unfortunately, the prolonged treatment of RLS using dopaminergic drugs, such as the approved pramipexole, can lead to a phenomenon called augmentation in which patients experience an increase in symptom severity, an earlier onset of symptoms during the night, the appearance of daytime symptoms, and/or the spread of symptoms to other parts of the body. Although, ropinirole is a dopamine agonist it appears to have a lower risk of augmentation and tolerance than other dopaminergic drugs, such as levodopa.

This study aims to evaluate effectiveness of the off-label use of ropinirole and gabapentin for the treatment of restless legs syndrome in patients on maintenance hemodialysis.

Hypothesis

Testing Superiority: The mean RLS symptom severity change in the ropinirole group is greater than placebo.

Testing Superiority: The mean RLS symptom severity change in the gabapentin group is greater than placebo.

Testing Equivalence: The mean RLS symptom severity change in the ropinirole group is within 10% of the gabapentin group.

Justification

Although these medications are considered first time pharmacologic treatment for patients with ESKD, few published studies provide treatment data for these patients. Treatment recommendations for this population are largely derived from extrapolation of data obtained in the general population, even though the pathophysiology for RLS in ESKD (termed "uremic RLS") may differ.

Restless legs syndrome is a chronic condition with fluctuating severity. The majority of the available published studies in the hemodialysis population were of short duration and small sample sizes. A six month intervention period will be used to evaluate the long-term effectiveness of ropinirole and gabapentin for the treatment of RLS symptoms in the hemodialysis population.

Primary Objectives

Evaluate the effectiveness of ropinirole and gabapentin on the severity of RLS symptoms in the hemodialysis population using the International Restless Legs Syndrome Study Group (IRLS) rating scale.

Secondary Objectives:

Evaluate the impact of ropinirole and gabapentin on the quality of life using the EQ-5D-5L is a two part standardized health status instrument.

Evaluate the impact of ropinirole and gabapentin on the quality of sleep using the Medical Outcomes Study Sleep Scale.

Evaluate the impact of ropinirole and gabapentin on the symptom burden using the Edmonton Symptom Assessment System Revised Renal.

Validate the addition of RLS and difficulty sleeping items on the Edmonton Symptom Assessment System Revised: Renal (ESAS-r: Renal).

Research Method/Procedures

Screening/Recruitment

A Nephrologist, Clinical Nurse Educator (CNE), and/or designate from the NARP, will identify patients meet the study criteria using minimal data from the Nephrology Information System (NIS). NIS is an electronic database used by NARP to record health for all patients in the program. Nephrologists and CNEs in the Northern Alberta Renal Program have access to the patient information in NIS as part of routine clinical care.

Initial contact with a potentially eligible participant will be made by an AHS NARP employee already involved in the clinical care of the patient, who will then determine the individual's willingness to be approached by the research study staff regarding participation and obtain their written consent to release their contact information to the researcher. The consent forms will be passed along to the researcher.

If the potential participant is agreeable a trained study coordinator will approach the eligible patient to introduce the study. The formal consent of a participant, using an HREB-approved consent form, will be obtained before that participant is submitted to any study intervention.

Potential participants will be advised (verbally and in written information) that participation is not required and refusal will not affect their health care or relationship with dialysis unit staff. Also, participants will be advised that they are free to leave the study at any time and would not be required to give a reason for withdrawal.

Potential participant initials will be used to track participants during recruitment so as not to approach the same patient multiple times. Recruitment information, such as reasons for refusal and date approached, will be recorded on Screening and Recruitment log.

Once eligible participants are recruited a baseline assessment will be completed and the participant will be randomized to the study groups. The participant will be instructed to start taking the study drug the same evening before bed. A follow up will be completed weekly for two months following the baseline date. Additional follow ups will occur at four and six months.

A total of 63 subjects will be enrolled and randomized into 3 groups: 23 participants will receive gabapentin, 23 participants will receive ropinirole, 17 participants will receive a placebo.

Study Design:

A six month, randomized, single-blind, placebo-controlled, parallel, multicenter, clinical trial comparing the effectiveness of ropinirole and gabapentin for the treatment of restless legs syndrome in patients on maintenance hemodialysis.

Intervention:

Once eligible participants are recruited a baseline assessment will be completed and the participant will be randomized to the study groups. The participant will be instructed to start taking the study drug the same evening before bed. A follow up will be completed weekly for two months following the baseline date to allow for monitoring and appropriate dose titration. Additional follow ups will occur at four and six months.

All patients treated with ropinirole will be started with a single dose of 0.25 mg once daily by mouth prior to bed as per the Alberta Kidney Care restless legs syndrome clinical guidelines used by the Northern Alberta Renal Program. Since the action of dopamine agonists generally starts 90 to 120 minutes after ingestion study participants will be instructed to take the ropinirole two hours before bed prior to symptom onset. Ropinirole may be taken with or without food. The ropinirole dose may be titrated upward in 0.25 mg increments every seven days as tolerated by the patient until symptom relief has been achieved or a maximum dose of 2.0 mg/day has been reached. In general, the effective dose for ropinirole is typically 2.0 mg or less and dosages higher than 2.0 mg have not been studied in the hemodialysis population.

All patients treated with gabapentin will be started with a single dose of 100mg once daily by mouth two hours prior to bed as per the Alberta Kidney Care restless legs syndrome clinical guidelines. Gabapentin may be taken with or without food. The dose may be increased in 100 mg increments every seven days as tolerated by the patient until symptom relief has been achieved or until a maximum study dose has been reached. As per the gabapentin product monograph dosing recommendations and current clinical RLS guidelines the maximum study gabapentin dose will 300 mg/day.

A placebo group will be used for comparison.

Plan for Data Analysis

The primary analysis will test changes in subject's IRLS scores between baseline and end of study (six month) follow up. Three separate analyses will be conducted, to test either superiority (gabapentin vs. placebo and ropinirole vs placebo), or equivalency (gabapentin vs. ropinirole). A t-test on the difference of means will be used for each superiority study; on the difference of mean percentage change for the equivalence study (with a set equivalence limit of 10%). For each treatment, a 50% decrease in IRLS scores from baseline will be considered clinically relevant, although a 30% decrease will be interpreted as a small improvement. An intent-to-treat (ITT) approach will be used in the primary analysis, although a per-protocol (PP) analysis will also be conducted for robustness.

Secondary analyses will test the mean change in subject's EQ-5D-5L quality of life scores, and MOS-SS sleep quality scales. Analyses on the differences between mean changes in scores will mirror those in the primary analysis. Analyses to validate the ESAS-r: Renal RLS and sleep quality measures will also be conducted. Criterion validity measured by Pearson correlation coefficient and multivariate regression analyses will be assessed using changes in IRLS scores to validate the RLS component, and changes in MOS-SS scores to validate the sleep quality component.

ELIGIBILITY:
Inclusion Criteria:

ESKD requiring hemodialysis

A symptom severity score of at least 4/10 on the restless legs ESAS-r: Renal question for two consecutive reporting periods (i.e over two months)

No RLS medication for two weeks prior to study period. Washout Period: Individuals that are receiving RLS medication but are still reporting a severity score of at least 4/10 on the restless legs ESAS-r: Renal they may be eligible if they discontinue their RLS medication for two weeks prior to baseline.

At least 18 years of age

Exclusion Criteria:

Dialysis vintage less than 3 months

Unstable medical conditions that prevents taking the study drugs or conditions that could affect efficacy treatment

Pregnancy

Previous adverse effects to gabapentin or ropinirole such as allergic reaction or augmentation

History of drug/alcohol abuse

Cognitive Impairment

Unable to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of ropinirole and gabapentin on the severity of RLS symptoms in the hemodialysis population. | up to 4 & 6 months after start of intervention.
  The International Restless Legs Syndrome Study Group (IRLS) rating scale was developed to measure the severity of RLS symptoms over the preceding seven days. The rating scale takes approximately 10 minutes to complete and consists of 10 questions rated from 0 - 4 (0 = none, 4 = very severe). The scale includes diagnostic features and questions to evaluate the intensity/frequency of RLS, associated sleep problems and impact of symptoms on mood and daily functioning. The total score ranges from 0 to 40; mild (1 - 10), moderate (11 - 20), severe (21 - 30) and very severe (31 - 40).

SECONDARY OUTCOMES:
Evaluate the impact of ropinirole and gabapentin on the quality of life. | EQ-5D-5L collected at baseline, and 1, 2, 4 & 6 months after start of intervention.
  The EQ-5D-5L is a two part standardized health status instrument used to measure quality of life over the previous four weeks. The questionnaire contains five, five-point Likert scale (1 = no problems, 5 = extreme problems) questions to evaluate mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The questionnaire also contains a 20 cm vertical visual analogue scale numbered 0 (worst health you can imagine) to 100 (best health you can imagine). This instrument is currently already in use within Alberta Health Services' (AHS) Northern Alberta Renal Program (NARP) for hemodialysis patients.
Evaluate the impact of ropinirole and gabapentin on the quality of sleep. | MOSS-SS collected at baseline, and 1, 2, 4 & 6 months after start of intervention.
  The Medical Outcomes Study Sleep Scale (MOS-SS) is used to evaluate six sleep parameter dimensions: sleep initiation, maintenance, respiratory problems quantity, perceived adequacy and somnolence over the past four weeks. Ten of the scale's 12 items are scored using a six-point Likert scale, one uses a five-point Likert scale, and one item is open-ended to record the average amount of hours slept. The scale takes less than five minutes to complete.
Evaluate the impact of ropinirole and gabapentin on the symptom burden. | The 10 item ESAS-r: Renal collected at baseline, and 1, 2, 4 & 6 months after start of intervention.
  The validated Edmonton Symptom Assessment System Revised Renal (ESAS-r: Renal) consists of 10 visual analogue scales with a superimposed zero to 10 severity scale for pain, activity, nausea, pruritus, depression, anxiety, drowsiness, appetite, well-being, and shortness of breath over the preceding 7 days. The scale for each symptom is anchored by the words 'No' and 'Severe' at zero and 10, respectively. Moderate intensity of any symptom is defined as 4 -6 and severe as 7 - 10 on the Likert scale. A total symptom distress score is calculated by summing of the scores for all 10 symptoms on the ESAS (ranges from 0 to 100).
Validate the addition of RLS and difficulty sleeping items on the Edmonton Symptom Assessment System Revised: Renal (ESAS-r: Renal). | The restless legs and difficulty sleeping items added to the ESAR-r: renal will be collected at baseline, and 1, 2, 4 & 6 months after start of intervention.
  The bi-monthly use of a modified 12 item ESAS-r: Renal has been implemented in to routine clinical care in Alberta Health Services' (AHS) Northern Alberta Renal Program (NARP) to assess patient symptom burden. The assessment used by clinicians includes two additional items scored from 0 to 10: sleep difficulties and restless legs. As a result of the additions, the total symptom distress score ranges from 0-120 for the ESAS version used in the NARP.

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Edmonton General Continuing Care Centre, Edmonton
  - Grey Nuns Community Hospital, Edmonton
  - Royal Alexandra Hospital, Edmonton
  - University of Alberta Hospital, Edmonton